

BiCRO-MO-010 Rev 2.0 22/03/2023

### STUDY PROTOCOL

### **TITLE**

SELF-CARE BEHAVIOURS OF TYPE 2 DIABETES MELLITUS PATIENTS:

A MULTICENTER PROSPECTIVE OBSERVATIONAL STUDY WITH 2 YEARS

**FOLLOW-UP** 

### **ACRONYM**

SCuDOS - Self-Care of Diabetes Observational Study

Version 1.1 - 29/11/2023

Status: Draft

#### **Study promoter**

University of Milan-Bicocca, Department of Medicine and Surgery

### Scientific director of the study

Prof. Davide Ausili - University of Milan-Bicocca

#### **Study authors**

Prof. Davide Ausili – University of Milan-Bicocca

Dr.ssa Michela Luciani – University of Milan-Bicocca

Dr.ssa Diletta Fabrizi – University of Milan-Bicocca

Prof Paola Rebora – University of Milan-Bicocca

Prof. Stefania Di Mauro – University of Milan-Bicocca

Dr. Rosario Caruso - Università degli studi di Milano, IRCCS Policlinico San Donato

Dr.sa Irene Baroni - IRCCS Policlinico San Donato

#### Statistician

Prof. Paola Rebora - University of Milan-Bicocca



BiCRO-MO-010 Rev 2.0 22/03/2023

### **Confidentiality statement**

This document contains confidential information belonging to University of Milano-Bicocca. Except as may be otherwise agreed to in writing, by accepting or reviewing these materials, you agree to hold such information in confidence and not to disclose it to others (except where required by applicable law), nor to use it for unauthorized purposes. In the event of actual or suspected breach of this obligation, Milano Bicocca University should be promptly notified.



BiCRO-MO-010 Rev 2.0 22/03/2023

# **Table of content**

| Background | 5 |
|---|---|
| Rationale | 5 |
| 1. Objectives and Indicators | 7 |
| 1.1 General Study Purpose | 7 |
| 1.1.1 Primary objective: | 7 |
| 1.1.2 Secondary objectives: | 7 |
| 1.2 Study Indicators | 8 |
| 1.2.1 Resource utilisation/health outcomes indicators | 8 |
| 1.2.2 Clinical Indicators | 8 |
| 1.2.3 Person-centred indicators | 9 |
| 1.2.4 Socio-demographic indicators. | 9 |
| 2. Study design | 9 |
| 3. Subject selection | 10 |
| 3.1 Inclusion criteria | 10 |
| 3.2 Exclusion criteria | 10 |
| 3.3 Sample size/Power evaluation | 10 |
| 3.4 Withdrawal | 11 |
| 4. Study procedures | 11 |
| 5. Data collection | 11 |
| 5.1. Short Form 12 - SF-12 (Italian, Version 1.0) | 12 |
| 5.2. Self-care of Diabetes Inventory - SCODI (Italian Version 1.0) | 13 |
| 5.3 EQ-5D-3L (Italian, Version 2) | 13 |
| 5.4 Problem Areas in Diabetes Questionnaire Short Form - PAID-5 (Italian) | 13 |
| 5.5 Pittsburgh Sleep Quality Index – PSQI (Italian) | 13 |
| 6. Data analysis | 14 |
| 7. Data integrity and quality assurance | 14 |
| 7.1 Monitoring and inspections | 14 |
| 7.2 Integrity of data collection | 15 |
| 7.3 Data Management | 15 |
| 7.4 Study documentation and storage | 15 |
| 7.5 Record keeping | 15 |
| 8. Ethical and legal aspects | 16 |
| 8.1 Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approval | 16 |



| 8.2 Protocol amendments | 16 |
|--------------------------------------|----|
| 8.3 Ethical Conduct of the Study | 17 |
| 8.4 Patient Information and Consent | 17 |
| 8.5 Privacy | 17 |
| 8.6 Insurance Policy | 18 |
| 8.7 Funding and conflict of interest | 18 |
| 9. Publication of Study Results | 18 |
| Attachment 1 – Schedule of events | 19 |
| Protocol Activities | 19 |
| References | 20 |



BiCRO-MO-010 Rev 2.0 22/03/2023

### Background

Chronic diseases represent a challenging issue for global health and constitute one of the main expenditures for healthcare organisations worldwide [1]. Patients' empowerment is considered a key principle in chronic illness management: available reports suggest that future health systems' sustainability will mainly depend on people's ability to manage their chronic conditions [2]. Chronically ill patients need to learn many specific behaviours in order to adhere to complex therapeutic regimes, to maintain their well-being and quality of life, to manage symptoms and to reduce disease complications [3]. All these behaviours, requiring knowledge, motivation, experience and skills, have been referred by many authors to the concept of self-care [4].

Self-care has been defined as "a process of maintaining health through health promoting practices and managing illness" [5, 6]. Key concepts of self-care of chronic diseases are self-care maintenance, self-care monitoring, and self-care management. Self-care maintenance comprises those behaviours used by patients with a chronic disease to maintain physical and emotional stability. Self-care monitoring refers to the process of observing oneself for changes in signs and symptoms. Self-care management includes those behaviours acted in response to signs and symptoms when they occur [6]. Several studies observed that self-care in chronic diseases improves quality of life, also reducing mortality and costs of healthcare services [7–9]. Although self-care is considered as a relevant intermediate outcome in chronic illness care, previous studies observed that chronically ill patients show low levels of self-care in recognising and managing their symptoms, in taking drug therapies, and in performing recommended behaviours [10–14].

### Rationale

Diabetes mellitus (DM) has been considered as one of the most serious chronic disease for morbidity and mortality all over the world [1, 15, 16]. It has been estimated that in 2019 the number



BiCRO-MO-010 Rev 2.0 22/03/2023

of persons affected by diabetes amounted to 463 million globally. Previsions showed that in 2045 the number will grow to about 700 million. DM accounted for 11.3% of global all-cause mortality among people aged between 20 to 79 years [15]. In Italy, about 5.3% of the population is affected by DM, for a total of 3.2 million people [17]. The prevalence of DM increases in older population and it has been estimated that diabetes will represent a real epidemic disease in the near future, impacting negatively on the health status of communities and the sustainability of health systems internationally [15, 18]. Type 2 diabetes mellitus (T2DM) accounts for more than 90% of diabetes cases [19], is associated with higher rate of cardiovascular disease [16], and leads to serious microvascular and macrovascular complications [15, 20, 21].

International scientific societies recognised self-care as a key factor for T2DM patients to maintain better health status and to avoid severe disease complications [21–24]. Self-care was shown to improve metabolic control [25, 26] and quality of life [27, 28] and to reduce cardiovascular risk [29], hospitalisations [30] and incidence of disease-related complications [31–33] in T2DM patients.

Although self-care has been recognised to be a crucial issue for people with T2DM, just a few studies were conducted in Italy to investigate patients' self-care behaviours, and their results need to be integrated by further research. In fact, some of the available studies used self-care measurement tools with several limitations [34, 35], as pointed out by systematic reviews [36, 37]. Further researches investigated self-care as one of the numerous study variables and the description of self-care behaviours was partial [38, 39]. Finally, many studies did not allow strong inferences about outcomes associated to self-care, because of their cross-sectional design or very short follow-up periods [12, 34, 39–41].

Measuring self-care, besides the benefits of standardisation, can help in better understanding the complexity and the dynamicity of the phenomenon in T2DM patients. The *Self-Care of Diabetes Inventory* (SCODI) has showed to be a valid and reliable tool to measure self-care maintenance, self-



BiCRO-MO-010 Rev 2.0 22/03/2023

care monitoring, and self-care management in the T2DM population [42, 43]. In these evaluations, HbA1c has a key role in clinical assessment of patient's metabolic control and it has also been validated as a surrogate endpoint of microvascular complications associated with diabetes [44–47].

Therefore, the present study could provide relevant information about the experience of people with T2DM, useful to better understand their self-care behaviours and to develop tailored healthcare interventions. Furthermore, study results could contribute to improve diabetes healthcare service organisation and to reduce disease-related costs. Details about study objectives, methods, tools, procedures and attended results will be described further on.

### 1. Objectives and Indicators

### 1.1 General Study Purpose

The general purpose of this study is to explore the experience of self-care in T2DM patients, to understand how to provide a higher quality assistance reducing complications and improving resource utilisation. The theoretical framework of the study will be the Middle-Range Theory of Self-Care of Chronic Illness, developed by Riegel and colleagues [6].

### 1.1.1 Primary objective:

- to estimate associations between self-care maintenance, self-care monitoring, and self-care management at baseline and HbA1c after a 12 months follow-up in T2DM patients;

### 1.1.2 Secondary objectives:

- to estimate associations between self-care maintenance, self-care monitoring, and self-care management at baseline and HbA1c after a 24 months follow-up in T2DM patients;
- to estimate associations between self-care maintenance, self-care monitoring, and self-care management and clinical outcomes (unplanned medical referral, access to emergency department, hospitalisation, indicators of metabolic control, incidence of diabetes complications, quality of life, death) over a 24 months years follow-up in T2DM patients.



## 

BiCRO-MO-010 Rev 2.0 22/03/2023

- to describe self-care maintenance, self-care monitoring, and self-care management and their directions over a 24 months follow-up in T2DM patients;
- to identify clinical and socio-demographic determinants of self-care maintenance, self-care monitoring, and self-care management in T2DM patients;
- to estimate the association between the trends of self-care maintenance, self-care monitoring, and self-care management and HbA1c over a 24 months follow-up;
- to integrate available data about validity and reliability of the SCODI;

### 1.2 Study Indicators

#### 1.2.1 Resource utilisation/health outcomes indicators

- Number of extra (both scheduled and unscheduled) diabetes medical or nursing referral (compared to the general planned routine) per year;
- Number of all-cause accesses to emergency departments per year;
- Number of all-cause hospitalisations per year;
- All-cause death;
- Participation to formal diabetes education programs during last year.

#### 1.2.2 Clinical Indicators

- Glycated haemoglobin (HbA1c);
- Time from the diagnosis of T2DM;
- Presence or absence and number of diabetes-related complications;
- Presence or absence and number of comorbidities;
- Ongoing medications and number of medications (including injections if patients are treated by insulin);
- Smoking habits;
- Lipid Profile (Total Cholesterol, HDL Cholesterol, LDL Cholesterol, Triglycerides);



BiCRO-MO-010 Rev 2.0 22/03/2023

- Liver Profile (ALT, AST, GGT);
- Renal Profile (Creatinine, estimated Glomerular Filtration Rate);
- Height, weight, and Body Mass Index (BMI);
- Arterial Blood Pressure and Heart Rate.

#### 1.2.3 Person-centred indicators

- Self-care maintenance (measured by the Self-Care of Diabetes Inventory, SCODI);
- Self-care monitoring (measured by the Self-Care of Diabetes Inventory, SCODI);
- Self-care management (measured by the Self-Care of Diabetes Inventory, SCODI);
- Self-care confidence (measured by the Self-Care of Diabetes Inventory, SCODI);
- Functional status (measured by the Short Form 12 questionnaire, SF12);
- Mental status (measured by the Short Form 12 questionnaire, SF12);
- Quality of life (measured by the EQ-5D-3L Quality of life Questionnaire);
- Diabetes-related distress (measured by the Problem Areas in Diabetes Questionnaire Short Form, PAID-5);
- Quality of sleep (measured by the Pittsburgh Sleep Quality Index, PSQI).

### 1.2.4 Socio-demographic indicators

- Age;
- Gender;
- Educational level;
- Job employment;
- Income level;
- Presence of formal or informal caregiver.

### 2. Study design

The study uses a multi-centred prospective observational design with 2 years follow-up.



BiCRO-MO-010 Rev 2.0 22/03/2023

### 3. Subject selection

Subjects will be contacted during their outpatient visit in Diabetes Centres and then asked to be enrolled in the study by investigators in a consecutive sequence, according to the following inclusion and exclusion criteria.

#### 3.1 Inclusion criteria

- Diagnosis of T2DM, as described in the available guidelines [49];
- Age over 18 years old;
- Adequate comprehension of Italian language;
- Signed and dated informed consent.

#### 3.2 Exclusion criteria

- Presence of documented psychiatric or neurodegenerative disease;
- Pregnancy;
- Any condition that, by the investigators' judgement, may limit adherence to study procedures.

  Disposition of subjects enrolled will be presented and their number at each visit will be tabulated.

  The reason for inclusion/exclusion will be tabulated and listed.

### 3.3 Sample size/Power evaluation

We expect to enrol around 300 patients who respect inclusion/exclusion criteria and are willing to participate to the study. An overall sample size of 300 subjects (of which 150 are expected to be at a low level of self-care monitoring) achieves 80% power at a 0.0500 significance level to detect a difference of about 0.4% (with a standard deviation of 1.1%) in HbA1c level between patient with lower and higher self-care monitoring after a follow-up of 12 months. This power takes into account a possible 20% of lost to follow-up. These assumptions are based on our preliminary data [42, 43] and consider a cut-off defining low and high level of self-care maintenance of 70/100 in a standardised

DEGLI STUDI

## STUDY PROTOCOL "SCuDOS" v. 1.1 (29.11.2023)

BiCRO-MO-010 Rev 2.0 22/03/2023

scale. The study has been sized on self-care monitoring, but similar results could be expected also in self-care maintenance and self-care management.

#### 3.4 Withdrawal

Patients may withdraw from the study at any time at their own request by withdrawing consent, or they may be withdrawn at any time at the discretion of the investigator for safety, behavioural, or administrative reasons. Every effort should be made to contact the patient for the follow-ups. In any circumstance, every effort should be made to document patient outcome, if possible.

### 4. Study procedures

Since the informed consent has been signed, socio-demographic and clinical data will be collected by medical records. At the beginning or at the end of the clinical standard outpatient visit, patients will be asked to complete study questionnaires. For the study procedures details, please refer to the schedule of events (Attachment 1).

### 5. Data collection

At the baseline (T<sub>0</sub>), socio-demographic and clinical data will be collected by medical records. Furthermore, five self-report questionnaires will be administered to participants.. Follow-up data, consisting of the same clinical data and questionnaires, will be collected by telephone at 12 (T<sub>1</sub>)and 24 months (T<sub>2</sub>). Moreover, intermediate follow-ups at 6 (T<sub>0.5</sub>) and 18 months (T<sub>1.5</sub>) will consist of the telephone administration of only 2 questionnaires. An overview of each timepoint data collection is shown in Figure 1, while the study procedures details are presented in the schedule of events (Attachment 1). For the questionnaires, short forms have been chosen to reduce the number of items and to improve respondent rates and adherence to protocol. All questionnaires were demonstrated to be valid and reliable, and they are widely used in research and clinical practice both at national and international level. Details about study questionnaires are reported below. All data will be recorded in eCRF..



BiCRO-MO-010 Rev 2.0 22/03/2023

The end of the study will be the date of conclusion of  $T_2$  data collection period, coinciding with 24 months (+ maximum 28 days) from the baseline ( $T_0$ ).

Figure 1. Data collection in each timepoint of the study



Notes: SF-12= Short Form 12; SCODI= Self-Care of Diabetes Inventory; EQ-5D-3L= EuroQol 5-Dimensions 3 Levels; PAID-5= Problem Areas in Diabetes Questionnaire Short Form; PSQI= Pittsburgh Sleep Quality Index.

### 5.1. Short Form 12 - SF-12 (Italian, Version 1.0)

This questionnaire is the short version of SF-36 and it has been chosen to evaluate the functional and mental well-being status. It is a validated tool, widely used, therefore it might help in data comparability. It has a 4 week retrospective span and inquires personal and social discomfort,



BiCRO-MO-010 Rev 2.0 22/03/2023

disabilities and self-description of the level of health perceived. It can be self-administered and it counts 12 items [51].

### 5.2. Self-care of Diabetes Inventory - SCODI (Italian Version 1.0)

This instrument has been developed by University of Milano-Bicocca and University of Pennsylvania grounded in Riegel Middle-Range Theory of Self-Care of Chronic Illness [6]. It can be self-administered and it counts 40 items. It is valid and reliable [42]. The SCODI questionnaire provides four measures: self-care maintenance, self-care monitoring, self-care management and self-care confidence. Each SCODI scale will provide a standardised 0-100 score. Higher scores mean better self-care.

#### 5.3 EQ-5D-3L (Italian, Version 2)

The EQ-5D-3L is a self-report tool, composed by a 5 items multiple questions section that investigate movement, hygiene, daily living activities tolerance, pain/discomfort and anxiety/depression. A Visual Analogue Scale is included in order to assess a general health status level as perceived by patients [52, 53].

### 5.4 Problem Areas in Diabetes Questionnaire Short Form - PAID-5 (Italian)

The PAID-5 is composed by 5 items and it can be self-administered. It has satisfactory sensitivity and specificity for recognition of diabetes-related emotional distress. The final score is between 0 and 100 points: a score higher than 40 points has been significantly associated to development of depression and other negative psychological outcomes [54].

#### 5.5 Pittsburgh Sleep Quality Index – PSOI (Italian)

The Pittsburgh Sleep Quality Index is a valid and reliable tool for assessing sleep quality [55, 56]. It comprises 19 items and it is self-administered. It provides a good and reliable differentiation between normal and pathological groups, with higher scores (cut-off 5 and higher) reported by people characterised by more impaired sleep quality [56].

DEGLI STUDI

## STUDY PROTOCOL "SCuDOS" v. 1.1 (29.11.2023)

BiCRO-MO-010 Rev 2.0 22/03/2023

### 6. Data analysis

Continuous data will be summarised with number of observations, mean value, standard deviation, median, quartiles, minimum, maximum, and 95% confidence intervals for the mean. Categorical data will be summarised by means of absolute and relative frequencies (counts and percentages).

Scores of SCODI's self-care scales will be standardised to 100 [42].

To estimate associations between self-care maintenance, self-care monitoring, and self-care management and HbA1c level at 12 months a t-test will be used.

The incidences of health and clinical outcomes over the follow-up will be computed by the Kaplan-Meier estimator in patients with low and high self-care at baseline (cut-off 70/100) and they will be compared by the log-rank test. The Cox model will be used to account for confounders. A Cox model will be also used to evaluate the impact of the SCODI (as continuous score) on health and clinical outcomes.

Self-care behaviours will be described by a boxplot and their relation with health and clinical outcomes over the whole follow-up will be modelled by longitudinal models.

Multiple linear regression analyses will be performed in order to identify clinical and sociodemographic determinants of self-care.

Explorative and confirmative factor analyses will be used to further evaluate the construct validity of the SCODI. Cronbach Alpha and further inter-item coefficients will be used to measure on a large sample the internal consistency of the tool.

### 7. Data integrity and quality assurance

### 7.1 Monitoring and inspections

The monitoring plan will comprise the site initiation visit, monitoring visits and the closure visit at the end of study by the study promoter. DEGLI STUDI

## STUDY PROTOCOL "SCuDOS" v. 1.1 (29.11.2023)

BiCRO-MO-010 Rev 2.0 22/03/2023

Institutional review board (IRB)/independent ethics committee (IEC) will have complete access to all the study documentation in case of inspection.

### 7.2 Integrity of data collection

Investigators must enter the information required by the protocol into the electronic Patient Data Collection Forms (eCRFs). Data entry will be a responsibility of the investigational site.

### 7.3 Data Management

Data Management is a responsibility of the promoter, which will supervise the study as quality control program.

Expert personnel will review the eCRFs for completeness and accuracy. Errors, omissions, or questions will be entered on data query forms, which will be returned to the investigational centre for resolution. After the investigator response is received by the data management centre, the resolutions will be entered into the database. A copy of the signed data query form will be kept with the print-out of the eCRFs by the investigational centre.

Appropriate measures, including encryption of data files containing person identifiable data, will be used to ensure confidentiality of patients' data.

### 7.4 Study documentation and storage

Data records must be kept for the maximum period permitted by the hospital or institution, and at least 15 years after the end of the study.

The investigator must agree to archive the documentation (this includes both electronic and paperbased records) of the study in an archive after completion or discontinuation of the study, if not otherwise notified.

The deletion process must ensure confidentiality of data and must be done in accordance with local requirements.

### 7.5 Record keeping

A DEGLI STUDI

## STUDY PROTOCOL "SCuDOS" v. 1.1 (29.11.2023)

BiCRO-MO-010 Rev 2.0 22/03/2023

To enable evaluations and/or audits from regulatory authorities, the investigator agrees to keep records, including the identity of all participating patients, their telephone numbers, all original signed informed consent forms, all CRFs, source documents, and adequate documentation of relevant correspondence. The records should be retained by the investigator according to the International Conference on Harmonisation (ICH), local regulations, or as specified in the Study Agreement. The encrypted file of the register containing patients' identities associated with their identification numbers and their telephone numbers will be sent to the promoter by tracked email, in order to allow the promoter to carry out telephone follow-ups. At the end of the telephone follow-ups, the file and the related emails will be destroyed by the promoter.

An electronic database will be created by the promoter and regular backup are assured.

At the end of the study, the database will be locked and a backup copy, saved on a non-rewritable CD, will be stored together with study documentation.

### 8. Ethical and legal aspects

### 8.1 Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approval

It is responsibility of the investigator to have prospective approval of the study protocol, protocol amendments, informed consent forms, and other relevant documents, if applicable, from the IRB/IEC. All correspondence with the IRB/IEC should be retained in the investigator file.

The principal investigator agrees to provide the IRB/IEC with all appropriate material, including a copy of the informed consent.

The study will not be initiated until the investigator obtains written approval of the research plan and the informed consent document from the appropriate IRB/IEC.

### 8.2 Protocol amendments

Every change in this protocol will be considered as an amendment and submitted prospectively to the IRB/IEC for approval.

DEGLI STUDI

STUDY PROTOCOL "SCuDOS" v. 1.1 (29.11.2023)

BiCRO-MO-010 Rev 2.0 22/03/2023

### 8.3 Ethical Conduct of the Study

The study will be conducted in accordance with legal and regulatory requirements, as well as the general principles set forth in the International Ethical Guidelines for Biomedical Research Involving Human Subjects [57], ICH Guidelines for Good Clinical Practice (GCP), and the Declaration of Helsinki [58].

### 8.4 Patient Information and Consent

All parties will ensure protection of patient personal data and will not include patient names on any sponsor forms, reports, publications, or in any other disclosures, except where required by laws. The informed consent form must be in compliance with ICH GCP, local regulatory requirements, and legal requirements.

The informed consent form used in this study, and any changes made during the course of the study, must be prospectively approved by the IRB/IEC before use.

The investigator must ensure that each study patient, or his/her legally acceptable representative, is fully informed about the nature and objectives of the study and possible risks associated with participation. The investigator, or a person designated by the investigator, will obtain written informed consent from each patient before any study-specific activity is performed. The investigator will retain the original of each patient's signed consent form.

### 8.5 Privacy

Regulatory authorities and/or IEC/IRB may request access to all source documents, data capture records, and other study documentation for one-site audit or inspection. Direct access to these documents must be guaranteed by the investigator, who must provide support at all times for these activities.

DEGLI STUDI

## STUDY PROTOCOL "SCuDOS" v. 1.1 (29.11.2023)

BiCRO-MO-010 Rev 2.0 22/03/2023

Data confidentiality will be maintained in all the phases of the study according to national and international regulation (European Union General Data Protection Regulation 2016/679 and amendments).

The patients' names will be asked by the promoter only for the telephone follow-up, as specified in the paragraph 7.5 Record keeping. A sequential identification number will be attributed to each patient enrolled in the study and to each centre. This number will identify the patient and must be included on all case report forms. In order to avoid identification errors, date of birth may also be reported on forms.

### 8.6 Insurance Policy

This is an observational study and patients are followed according to usual clinical practice, with the exception of the completion of questionnaires and the participation of interviews. No specific insurance is required for the study.

### 8.7 Funding and conflict of interest

No funding are allocated for this study. If a possibility to get funded arise before completion of the study, the project will be submitted for funding and an amendment will be presented to the IEC/IRB. No conflict of interest to be declared.

### 9. Publication of Study Results

All data produced are property of study promoters (in the legal person of Professor Davide Ausili – University of Milano-Bicocca) and will be made public after all data have been analysed and the study results are available. Eventual publications using single centre data will be prospectively agreed with the promoter and, in any case study promoters will be involved in the manuscript authorship.



BiCRO-MO-010 Rev 2.0 22/03/2023

# **Attachment 1 – Schedule of events**

| Protocol Activities | T <sub>0</sub><br>Baseline | T <sub>0.5</sub> Month 6 ± 28 days | T <sub>1</sub> Month 12 ± 28 days | T <sub>1.5</sub> Month 18 ± 28 days | T <sub>2</sub> Month 24 ± 28 days |
|---|---|---|---|---|---|
| BASELINE DOCUMENTATION | | | | | |
| Informed consent No activity should be performed before obtaining signed and dated informed consent | х | | | | |
| Review of inclusion and exclusion criteria by the researcher | х | | | | |
| Disease history Assess diabetes history, diabetes-related medications and complications, co- morbidities, ongoing drugs, smoking habits. | x | | x | | x |
| Physical assessment Height (at screening only), weight, abdominal circumference, BMI, blood pressure and pulse rate | х | | x | | x |
| LABORATORY STUDIES | | | | | |
| HbA1c (mmol and %) | X | | X | | X |
| Lipidic profile Total Cholesterol, HDL Cholesterol, LDL Cholesterol, Triglycerides | X | | X | | X |
| Renal and Liver profile Creatinine, estimated GFR, ALT, AST, GGT | X | | X | | X |
| QUESTIONNAIRES | | | | | |
| Short Form 12 (SF-12) | X | | X | | X |
| Self-Care of Diabetes Inventory (SCODI) | X | Х | X | х | X |
| Quality of Life (EQ-5D-3L) | X | Х | X | х | X |
| Problem Areas in Diabetes Questionnaire<br>Short Form (PAID-5) | х | | x | | х |
| Pittsburgh Sleep Quality Index (PSQI) | X | | X | | x |
| OTHER ASSESSMENT | | | | | |
| Events Any referral or unplanned diabetes visit, request for home care assistance, hospitalisation, access to emergency care, | х | | х | | x |



BiCRO-MO-010 Rev 2.0 22/03/2023

| death, received diabetes education in the |
|-------------------------------------------|
| last year. |

### References

- 1. World Health Organization (2018) Noncommunicable Diseases Report 2018. Geneva
- 2. Prince MJ, Wu F, Guo Y, et al (2015) The burden of disease in older people and implications for health policy and practice. Lancet 385:549–562
- 3. Riegel B, Dunbar SB, Fitzsimons D, et al (2019) Self-care research: Where are we now?

  Where are we going? Int J Nurs Stud 103402. https://doi.org/10.1016/j.ijnurstu.2019.103402
- 4. Lommi M, Matarese M, Alvaro R, et al [The evolution of the concept of self-care in the healthcare system: a narrative literature review]. Prof Inferm 68:155–66. https://doi.org/10.7429/pi.2015.682155
- 6. Riegel B, Jaarsma T, Strömberg A (2012) A Middle-Range Theory of Self-Care of Chronic Illness. Adv Nurs Sci 35:194–204. https://doi.org/10.1097/ANS.0b013e318261b1ba
- 7. Rochfort A, Beirne S, Doran G, et al (2018) Does patient self-management education of primary care professionals improve patient outcomes: A systematic review. BMC Fam Pract 19:. https://doi.org/10.1186/s12875-018-0847-x
- 8. Darkins A, Kendall S, Edmonson E, et al (2015) Reduced cost and mortality using home telehealth to promote self-management of complex chronic conditions: a retrospective matched cohort study of 4,999 veteran patients. Telemed J E Health 21:70–6. https://doi.org/10.1089/tmj.2014.0067
- 9. Hamar GB, Rula EY, Coberley C, et al (2015) Long-term impact of a chronic disease



BiCRO-MO-010 Rev 2.0 22/03/2023

management program on hospital utilization and cost in an Australian population with heart disease or diabetes. BMC Health Serv Res 15:174. https://doi.org/10.1186/s12913-015-0834-z

- Cocchieri A, Riegel B, D'Agostino F, et al (2015) Describing self-care in Italian adults with heart failure and identifying determinants of poor self-care. Eur J Cardiovasc Nurs 14:126– 36. https://doi.org/10.1177/1474515113518443
- 11. Buck HG, Dickson VV, Fida R, et al (2015) Predictors of hospitalization and quality of life in heart failure: A model of comorbidity, self-efficacy and self-care. Int J Nurs Stud 52:1714–22. https://doi.org/10.1016/j.ijnurstu.2015.06.018
- 12. Nicolucci A, Kovacs Burns K, Holt RIG, et al (2013) Diabetes Attitudes, Wishes and Needs second study (DAWN2<sup>TM</sup>): Cross-national benchmarking of diabetes-related psychosocial outcomes for people with diabetes. Diabet Med 30:767–777. https://doi.org/10.1111/dme.12245
- 13. Crowley MJ, Holleman R, Klamerus ML, et al (2014) Factors associated with persistent poorly controlled diabetes mellitus: clues to improving management in patients with resistant poor control. Chronic Illn 10:291–302. https://doi.org/10.1177/1742395314523653
- 14. Caro-Bautista J, Martín-Santos FJ, Villa-Estrada F, et al (2015) Using qualitative methods in developing an instrument to identify barriers to self-care among persons with type 2 diabetes mellitus. J Clin Nurs 24:1024–37. https://doi.org/10.1111/jocn.12740
- 15. International Diabetes Federation (2019) IDF Diabetes Atlas 9th Edition. Brussels
- 16. World Health Organization (2016) Global Report on Diabetes. Geneva
- 17. Istituto Nazionale di Statistica (2017) Diabetes in Italy. Rome
- 18. Zhou B, Lu Y, Hajifathalian K, et al (2016) Worldwide trends in diabetes since 1980: a pooled analysis of 751 population-based studies with 4·4 million participants. Lancet



- 387:1513–1530. https://doi.org/10.1016/S0140-6736(16)00618-8
- Chatterjee S, Khunti K, Davies MJ (2017) Type 2 diabetes. Lancet 389:2239–2251.
   https://doi.org/10.1016/S0140-6736(17)30058-2
- Fowler MJ (2008) Microvascular and Macrovascular Complications of Diabetes. Clin Diabetes 26:77–82. https://doi.org/10.2337/diaclin.26.2.77
- American Association of Diabetes Educators (2009) AADE Guidelines for the Practice of Diabetes Self-Management Education and Training (DSME/T). Diabetes Educ 35:85S-107S. https://doi.org/10.1177/0145721709352436
- 22. Powers MA, Bardsley J, Cypress M, et al (2016) Diabetes Self-management Education and Support in Type 2 Diabetes: A Joint Position Statement of the American Diabetes Association, the American Association of Diabetes Educators, and the Academy of Nutrition and Dietetics. Clin Diabetes 34:70–80. https://doi.org/10.2337/diaclin.34.2.70
- American Diabetes Association (2019) Standards of Medical Care in Diabetes-2019.
   Diabetes Care 42:S1–S193. https://doi.org/10.2337/dc19-Sint01
- 24. Felton A-M, Hall M (2015) Diabetes in Europe policy puzzle: the state we are in. Int Diabetes Nurs 12:3–7. https://doi.org/10.1179/2057331615z.0000000007
- 25. Yuan C, Lai CWK, Chan LWC, et al (2014) The Effect of Diabetes Self-Management Education on Body Weight, Glycemic Control, and Other Metabolic Markers in Patients with Type 2 Diabetes Mellitus. J Diabetes Res 2014:1–6. https://doi.org/10.1155/2014/789761
- 26. Walker RJ, Smalls BL, Hernandez-Tejada MA, et al (2014) Effect of diabetes self-efficacy on glycemic control, medication adherence, self-care behaviors, and quality of life in a predominantly low-income, minority population. Ethn Dis 24:349–355
- 27. Kargar Jahromi M, Ramezanli S, Taheri L (2014) Effectiveness of diabetes self-management education on quality of life in diabetic elderly females. Glob J Health Sci 7:10–5.



BiCRO-MO-010 Rev 2.0 22/03/2023

https://doi.org/10.5539/gjhs.v7n1p10

- 28. Chao J, Yang L, Xu H, et al (2015) The effect of integrated health management model on the health of older adults with diabetes in a randomized controlled trial. Arch Gerontol Geriatr 60:82–88. https://doi.org/10.1016/j.archger.2014.10.006
- 29. Sicuro J, Charrier L, Berchialla P, et al (2014) Self-management education by group care reduces cardiovascular risk in patients with type 2 diabetes: analysis of the ROMEO clinical trial. Diabetes Care 37:e192-3. https://doi.org/10.2337/dc14-1054
- 30. Adepoju OE, Bolin JN, Phillips CD, et al (2014) Effects of diabetes self-management programs on time-to-hospitalization among patients with type 2 diabetes: A survival analysis model. Patient Educ Couns 95:111–117. https://doi.org/10.1016/j.pec.2014.01.001
- 31. Williams IC, Utz SW, Hinton I, et al (2014) Enhancing Diabetes Self-care Among Rural African Americans With Diabetes: Results of a Two-year Culturally Tailored Intervention.

  Diabetes Educ 40:231–239. https://doi.org/10.1177/0145721713520570
- 32. Shreck E, Gonzalez JS, Cohen HW, Walker EA (2014) Risk perception and self-management in urban, diverse adults with type 2 diabetes: the improving diabetes outcomes study. Int J Behav Med 21:88–98. https://doi.org/10.1007/s12529-013-9291-4
- 33. Shrivastava SR, Shrivastava PS, Ramasamy J (2013) Role of self-care in management of diabetes mellitus. J. Diabetes Metab. Disord. 12
- 34. Ausili D, Bezze S, Canizzaro C, et al (2015) Self-care assessment in type-2 diabetes: the Italian translation and validation of the Summary of Diabetes Self-Care Activities. Prof Inferm 68:9–18. https://doi.org/10.7429/pi.2015.681009
- 35. Bagnasco A, Di Giacomo P, Da Rin Della Mora R, et al (2014) Factors influencing self-management in patients with type 2 diabetes: a quantitative systematic review protocol. J Adv Nurs 70:187–200. https://doi.org/10.1111/jan.12178



## 

- 36. Lu Y, Xu J, Zhao W, Han H-R (2016) Measuring Self-Care in Persons With Type 2 Diabetes: A Systematic Review. Eval Health Prof 39:131–84. https://doi.org/10.1177/0163278715588927
- 37. Caro-Bautista J, Martín-Santos FJ, Morales-Asencio JM (2014) Systematic review of the psychometric properties and theoretical grounding of instruments evaluating self-care in people with type 2 Diabetes Mellitus. J Adv Nurs 70:1209–1227. https://doi.org/10.1111/jan.12298
- 38. Nicolucci A, Rossi MC, Pellegrini F, et al (2014) Benchmarking network for clinical and humanistic outcomes in diabetes (BENCH-D) study: Protocol, tools, and population.

  Springerplus 3:1–9. https://doi.org/10.1186/2193-1801-3-83
- 39. Peyrot M, Burns KK, Davies M, et al (2013) Diabetes Attitudes Wishes and Needs 2 (DAWN2): a multinational, multi-stakeholder study of psychosocial issues in diabetes and person-centred diabetes care. Diabetes Res Clin Pract 99:174–84. https://doi.org/10.1016/j.diabres.2012.11.016
- 40. Holt RIG, Nicolucci A, Kovacs Burns K, et al (2013) Diabetes Attitudes, Wishes and Needs second study (DAWN2<sup>TM</sup>): cross-national comparisons on barriers and resources for optimal care--healthcare professional perspective. Diabet Med 30:789–98. https://doi.org/10.1111/dme.12242
- 41. Kovacs Burns K, Nicolucci A, Holt RIG, et al (2013) Diabetes Attitudes, Wishes and Needs second study (DAWN2<sup>TM</sup>): cross-national benchmarking indicators for family members living with people with diabetes. Diabet Med 30:778–88. https://doi.org/10.1111/dme.12239
- 42. Ausili D, Barbaranelli C, Rossi E, et al (2017) Development and psychometric testing of a theory-based tool to measure self-care in diabetes patients: the Self-Care of Diabetes Inventory. BMC Endocr Disord 17:66. https://doi.org/10.1186/s12902-017-0218-y



50.

## 

- 43. Ausili D, Rossi E, Rebora P, et al (2018) Socio-demographic and clinical determinants of self-care in adults with type 2 diabetes: a multicentre observational study. Acta Diabetol 55:691–702. https://doi.org/10.1007/s00592-018-1135-x
- 44. Sherwani SI, Khan HA, Ekhzaimy A, et al (2016) Significance of HbA1c Test in Diagnosis and Prognosis of Diabetic Patients. Biomark Insights 11:95–104.
  https://doi.org/10.4137/BMI.S38440
- 45. American Diabetes Association AD (2019) 6. Glycemic Targets: Standards of Medical Care in Diabetes-2019. Diabetes Care 42:S61–S70. https://doi.org/10.2337/dc19-S006
- 46. Schnell O, Alawi H, Battelino T, et al (2013) Self-monitoring of blood glucose in type 2 diabetes: recent studies. J Diabetes Sci Technol 7:478–88.
  https://doi.org/10.1177/193229681300700225
- 47. Cagney DN, Sul J, Huang RY, et al (2018) The FDA NIH Biomarkers, EndpointS, and other Tools (BEST) resource in neuro-oncology. Neuro Oncol 20:1162–1172. https://doi.org/10.1093/neuonc/nox242
- 48. Thorne SE (2016) Interpretive description : qualitative research for applied practice, 2nd ed.

  Routledge, New York and London
- 49. Associazione Medici Diabetologi, Società Italiana di Diabetologia (2018) Standard italiani per la cura del diabete mellito 2018
- 51. Ware JE, Kosinski M, Keller SD (1996) A 12-Item Short-Form Health Survey: Construction of Scales and Preliminary Tests of Reliability and Validity. Med Care 34:220–233. https://doi.org/10.1097/00005650-199603000-00003
- 52. Rabin R, De Charro F (2001) EQ-5D: A measure of health status from the EuroQol Group.In: Annals of Medicine. Royal Society of Medicine Press Ltd, pp 337–343



- 53. Savoia E, Fantini MP, Pandolfi PP, et al (2006) Assessing the construct validity of the Italian version of the EQ-5D: Preliminary results from a cross-sectional study in North Italy. Health Qual Life Outcomes 4:. https://doi.org/10.1186/1477-7525-4-47
- 54. McGuire BE, Morrison TG, Hermanns N, et al (2010) Short-form measures of diabetes-related emotional distress: The Problem Areas in Diabetes Scale (PAID)-5 and PAID-1. Diabetologia 53:66–69. https://doi.org/10.1007/s00125-009-1559-5
- 55. Buysse DJ, Reynolds CF, Monk TH, et al (1989) The Pittsburgh sleep quality index: A new instrument for psychiatric practice and research. Psychiatry Res 28:193–213. https://doi.org/10.1016/0165-1781(89)90047-4
- 56. Curcio G, Tempesta D, Scarlata S, et al (2013) Validity of the Italian version of the Pittsburgh Sleep Quality Index (PSQI). Neurol Sci 34:511–9. https://doi.org/10.1007/s10072-012-1085-y
- 57. Council for International Organizations of Medical Sciences (2002) International Ethical Guidelines for Biomedical Research Involving Human Subjects - CIOMS. CIOMS Publications
- 58. World Medical Association (2013) World Medical Association Declaration of Helsinki:
  Ethical Principles for Medical Research Involving Human Subjects. JAMA 310:2191–2194.
  https://doi.org/10.1001/jama.2013.281053